CLINICAL TRIAL: NCT05135910
Title: An Open Label Phase 2a Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of Hallux Terbinafine Subungual Gel Administered to the Toenail Bed of Patients With Distal-Lateral Subungual Onychomycosis
Brief Title: To Evaluate Hallux Terbinafine Subungual Gel (HSG) in the Treatment of Onychomycosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hallux, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSG-201
Record Dates: First submitted 2021-10-28; First posted 2021-11-26 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Onychomycosis of Toenail
Keywords: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HSG (Experimental): Hallux terbinafine subungual gel
  Interventions: Drug: Hallux Terbinafine Subungual Gel

INTERVENTIONS:
Drug: Hallux Terbinafine Subungual Gel — Hallux Terbinafine Subungual Gel (HSG) administered every 1 to 2 months over 44 weeks.
  Other Names: HSG

SUMMARY:
The key objective is to establish the efficacy, safety, tolerability, and pharmacokinetics of investigational drug Hallux Terbinafine Subungual Gel (HSG) administered over 44 weeks to patients with distal-lateral subungual onychomycosis (DLSO).

DETAILED DESCRIPTION:
Primary Efficacy: To identify patients achieving Complete Cure in the target toenail at Week 52.

Secondary Efficacy: To identify patients that have achieved 1) Clinical Cure, 2) Mycological Cure, and/or 3) Positive Response in the target toenail at Week 52.

Plasma Pharmacokinetics: To characterize concentrations of terbinafine and major metabolite in a subpopulation of patients over the study period.

Nail Pharmacokinetics: To characterize concentrations of terbinafine and major metabolite in distal nail clippings in patients over the study period.

HSG Safety and Tolerability Profile: To establish from plasma pharmacokinetics, related adverse events, treatment site reactions, pain, clinically significant changes in medical condition and/or medications, and clinically significant changes in liver function, serum chemistry, urinalysis, and complete blood count over the study period.

Subungual Topical Procedure: To establish the ease and durability of once monthly and once bi-monthly HSG subungual topical treatments, the Investigator will record at selected time points 1) nail measurements indicating progressive clearing, 2) the ease and depth of each topical administration, 3) the investigational drug volume administered each treatment, and 4) patient tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 18 - 75 years of age inclusive
* Patients with DLSO of at least one great toe
* Patients with DLSO in the target toe confirmed by positive KOH and positive fungal culture for dermatophytes
* Willingness to abstain from pedicures, nail clipping, or application of nail polish or nail cosmetics to their toenails over the study period

Exclusion Criteria:

* History of any significant chronic fungal disease other than onychomycosis or an immunocompromised condition
* Any previous surgery to or abnormalities of the target toe that in the investigator's opinion could prevent the toenail surface area from clearing even if eradication of the DLSO infection is achieved
* Participation in another clinical study of an investigational drug or device within 3 months of screening
* No administration of oral terbinafine or another oral antifungal within 6 months of screening
* No topical antifungal used for onychomycosis or a dermatophyte infection (i.e. tinea pedis) within 3 months of screening
* No uncontrolled diabetes mellitus
* No severe psoriasis or severe atopic dermatitis

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete Cure at Week 52 in the Target Toe | Week 52
  Complete Cure is defined as 1) 100% healthy, clear nail, and 2) negative mycology. Healthy, clear nail is absent any disease involvement attributable to DLSO and is determined by Investigator Global Assessment (IGA). Negative mycology is defined as zero visualization of septate hyphae by KOH microscopy (negative KOH) combined with a fungal culture negative for causal dermatophytes (negative fungal culture).

SECONDARY OUTCOMES:
Clinical Cure in the Target Toe | Week 52
  100% healthy, clear nail
Mycological Cure in the Target Toe | Week 52
  Negative KOH, negative fungal culture
Positive Response in the Target Toe | Week 52
  ≥ 80% decrease in disease involvement

OTHER OUTCOMES:
Plasma Pharmacokinetics | Week 52
  To characterize plasma concentrations of terbinafine and metabolite from a subset of patients over the study period
Nail Pharmacokinetics | Week 52
  To characterize nail concentrations of terbinafine and metabolite from patients over the study period
Subungual Topical Procedure | Week 44
  To evaluate the ease and durability of once monthly and once bi-monthly HSG subungual topical treatments to the target toe over 44 weeks. Nail measurements indicating progressive clearing are recorded from an Investigator Global Assessment scale referencing % disease involvement corroborated by nail image analysis. The ease and durability of subungual topical treatment is established using a 5-point Likert Scale. Patient local tolerability is established using a Treatment Site Assessment Scale and Pain Intensity Scale.
Patient Global Assessment | Week 52
  To establish each patient's impression of DLSO improvement in their target toe over the study period, patients will reference the following scale (0 = clear of DLSO, 1 = marked improvement of DLSO, 2 = moderately improved DLSO, 3 = slightly improved DLSO, 4 = unchanged, 5 = worse)
Safety and Tolerability: Established from patient incidence of Treatment-Emergent Adverse Events | Monitored from screening visit to end of study visit (Week 52)
  Indicated by the number of patients with treatment-related adverse events assessed by Common Terminology Criteria for Adverse Events (CTCAE)
Safety and Tolerability: Established from clinical laboratory results | Monitored at selected time points from screening visit to end of study visit (Week 52)
  Indicated by clinically significant changes in patient liver function, serum chemistry, urinalysis, and complete blood count over the study period
Safety and Tolerability: Established from patient reported medical condition and use of medications | Monitored from screening visit to end of study visit (Week 52)
  Monitored by assessing clinically significant changes in patient medical condition and/or use of medications over the study period

CONTACTS AND LOCATIONS:
Overall Officials: Lewis H. Freed, DPM, Principal Investigator — OrthoArizona, East Valley Foot & Ankle Specialists; Terry M. Jones, MD, Principal Investigator — J&S Studies; Daniel P. Mallett, DPM, Principal Investigator — Front Range Foot and Ankle Clinic; Phoebe Rich, MD, Principal Investigator — Oregon Dermatology and Research Center
Locations (4):
- United States (4):
  - OrthoArizona - East Valley Foot & Ankle Specialists, Mesa, Arizona
  - Front Range Foot and Ankle Clinic, Parker, Colorado
  - Oregon Dermatology & Research Center, Portland, Oregon
  - J&S Studies, College Station, Texas

IPD SHARING:
Plan to Share IPD: No
This is a phase II study. Individual participant data (IPD) of this study will not be shared.